CLINICAL TRIAL: NCT04837560
Title: Safety and Efficacy of the ElastiMed's SACS 2.0 - Smart Active Compression Stocking
Brief Title: Safety and Efficacy of the ElastiMed's SACS 2.0 - Smart Active Compression Stocking for the Treatment of Venous Edema
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ElastiMed ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-002
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Edema Leg; Compression; Vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporarily or permanently wheelchair users which suffer from Venous Edema (Experimental): Temporarily or permanently wheelchair users which suffer from Venous Edema
  Interventions: Device: ElastiMed's SACS 2.0

INTERVENTIONS:
Device: ElastiMed's SACS 2.0 — A wearable medical device that improve circulation using smart materials

SUMMARY:
Device Efficacy:

The primary efficacy assessment will be defined as successful if the edema volume will be reduced over time after using the SACS 2.0 device.

Treatment and edema evaluation will be performed in comparison to a standard compression bandage. The treatment will be performed for several hours during the subject's daily rest time.

The Measurements will be performed daily before treatment initiation and without the device on the leg (baseline) (T0); and after four hours of device operation.

The edema volume will be measured by a calf circumference measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 to 80 years old
2. Venous edema patients diagnosed by an indent in the skin following finger pressure.
3. Venous edema in both calves
4. Temporarily or permanently wheelchair users which are expected to remain so according to the investigator's discretion
5. Subjects able to provide a written informed consent
6. No existence of DVT according to leg deep vein Duplex test

Exclusion Criteria as reported by patients: :

1. Positive pregnancy test
2. Breastfeeding woman
3. moderate or severe Congestive heart failure
4. Cellulitis of tissues of the lower limb.
5. Infectious Dermatitis of the lower limb
6. Acute or within 6 weeks of a deep vein thrombosis (DVT).
7. Postphlebetic patients
8. Known hypersensitivity to any component of the device
9. Subjects unable to provide informed consent
10. Active cancer at the root of the limb or in the adjacent quadrant
11. Any limitation of renal function- according to the investigator's discretion
12. Any limitation of liver function - according to the investigator's discretion
13. Subject who cannot commit to a month of intensive standard therapy
14. Wound or other skin condition that, according to the investigator's discretion, might be aggravated by the garment
15. Currently participating in another clinical trial or have completed their participation in a clinical trial within 30 days of screening
16. Other physical and/or mental conditions that, according to the investigator's discretion, prevent the subject from participating in the trial and completing its assessments
17. Cardiac or cerebral pacemaker or stimulator
18. Patients after orthopedic / vascular injury in the lower extremities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | Device operation hours during 10 business days
  Accumulative rate of device related SAEs throughout the trial duration.
Efficacy Endpoint | Device operation hours during 10 business days
  To demonstrate the efficacy by following the edema volume reduction after device application, in venous edema subjects, by measuring the calf circumference

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | Device operation hours during 10 business days
  To demonstrate the efficacy by changing the edema volume after using the SACS 2.0 device at least as much as after using a compression bandage

CONTACTS AND LOCATIONS:
Overall Officials: Israel Dudkiewicz, Prof., Principal Investigator — Sheba Medical Center at Tel HaShomer
Locations (1):
- Sheba Medical Center at Tel HaShomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No